CLINICAL TRIAL: NCT06389383
Title: Pilot Study - Monitoring the Nasal Microbiome and Viral Respiratory Infections in Newborn Hospitalized in Neonatalogy. Metatranscriptomic Approach by New Generation Sequencing From High Respiratory Swabs.
Brief Title: Pilot Study - Monitoring the Nasal Microbiome and Viral Respiratory Infections in Newborn Hospitalized in Neonatalogy.
Acronym: NEONATMICROBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-0182
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Newborn; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nasal swab (Other): * Nasal swab once a week for the duration of the stay in intensive care unit/intensive care (procedure already carried out routinely to detect nasal staphylococcus once a week).
  * Nasal swab every 14 days when the newborn is hospitalized in routine care/kangaroo unit/hospitalization at home
  Interventions: Other: Nasal Swab

INTERVENTIONS:
Other: Nasal Swab — * Nasal swab once a week for the duration of the stay in intensive care unit/intensive care (procedure already carried out routinely to detect nasal staphylococcus once a week).
  * Nasal swab every 14 days when the newborn is hospitalized in routine care/kangaroo unit/hospitalization at home

SUMMARY:
The objective of our study is therefore to study the evolution of the respiratory microbiome of hospitalized newborns, its interaction with viral infections and their impacts on the evolution of newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborn hospitalized in intensive care or neonatal intensive care.
* Whose parents were able to be informed of the study and who signed consent.
* Parents affiliate to the social security system

Exclusion Criteria:

* Refusal of parental consent
* Parents who are minors or under guardianship, curatorship, safeguard of justice or legal protection.
* Newborn having already left the hospital/returned home before inclusion
* Hospitalization beyond the first 48 hours of life
* Only palliative care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
rate of viral infections | from baseline to end of hospitalization (up to 2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France